CLINICAL TRIAL: NCT01060813
Title: Study of the Benefit of Exercise and Aminoacid Supplements in Cirrhotic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, German Soriano, Dr. German Soriano Pastor, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-AMI-2009-17
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2011-09

CONDITIONS: Cirrhosis
Keywords: cirrhosis; exercise; leucin; glutamine synthetase
MeSH Terms: conditions — Fibrosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise + Leucine (Active Comparator): Patients will receive leucine 10 g/d po + exercise for 3 months
  Interventions: Dietary Supplement: Leucine supplements
- Leucine without exercise (Active Comparator): patients will receive leucine 10 g/d po
  Interventions: Dietary Supplement: Leucine supplements

INTERVENTIONS:
Dietary Supplement: Leucine supplements — leucine supplements
  Other Names: No other names

SUMMARY:
This is a pilot study including 20 cirrhotic patients that will be randomized to receive during 3 months leucine vs leucine plus a programme of physical exercise specially designed for cirrhotic patients. The hypothesis is that physical exercise in cirrhotic patients could increase muscle mass (and therefore glutamine synthetase activity leading to a higher blood ammonium clearance) and quality of life. Safety of physical exercise in cirrhotic patients will be strictly assessed.

ELIGIBILITY:
Inclusion Criteria:

* compensated liver cirrhosis.

Exclusion Criteria:

* hepatocellular carcinoma,
* active alcoholism (less than 1 year),
* decompensated cirrhosis,
* variceal bleeding less than 3 months,
* contraindication for exercise.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
glutamine synthetase activity | three months

SECONDARY OUTCOMES:
quality of life | three months

CONTACTS AND LOCATIONS:
Overall Officials: German Soriano, MD, PhD, Principal Investigator — Department of Gastroenterology, Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain